CLINICAL TRIAL: NCT06802718
Title: A Prospective Randomized Controlled Trial of Interferon-alpha As Maintenance Therapy for Favorable-risk Acute Myeloid Leukemia
Brief Title: Interferon-alpha As Maintenance Therapy for Favorable-risk Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHD001-001
Record Dates: First submitted 2024-12-21; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interferon Group (Experimental): Polyethylene glycol interferon alpha-2b injection 135 μg/week was subcutaneously given for 6 months.
  Interventions: Drug: Interferon
- Control Group (No Intervention): Observational follow-up without receiving any maintenance treatment.

INTERVENTIONS:
Drug: Interferon — Polyethylene glycol interferon alpha-2b injection 135 μg/week was subcutaneously given for 6 months.
  Arms: Interferon Group

SUMMARY:
This research focuses on a prospective, randomized, controlled trial of "Interferon-alpha as maintenance therapy for favorable-risk acute myeloid leukemia." By fully utilizing prospective, randomized, controlled clinical trial and studying the negative conversion of MRD and the survival of favorable-risk AML patients, it aims to explore the efficacy and safety of Interferon-alpha in the maintenance treatment of favorable-risk AML and identify effective measures to prevent relapse, thereby improving the survival of favorable-risk AML patients. The primary endpoint is the negative conversion of MRD at 6 months. The secondary endpoints include the 2-year cumulative incidence of relapse, 2-year event-free survival (EFS), 2-year overall survival (OS), and safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old (including 18 and 70 years old) with newly diagnosed favorable-risk AML (2022 ELN risk group classification).
* Achieved CR1 after 1-2 cycles of standard chemotherapy.
* Completed 4-6 cycles of consolidation chemotherapy (including at least 2 cycles of high-dose Cytarabine HDAC regimem).
* At the end of consolidation treatment, bone marrow examination confirmed in CR1, flow cytometry MRD negative, but molecular MRD genes (RUNX1:: RUNX1T1, NPM1, and CBFb:: MYH11) decreased by > 3 log, but still detectable.
* Performance status score of 0-2 (ECOG).
* Liver function: ALT and AST ≤ 2.5 times the upper limit of normal, bilirubin ≤ 2 times the upper limit of normal.
* Kidney function: Creatinine ≤ 1.5 times the upper limit of normal.

Exclusion Criteria:

* Acute promyelocytic leukemia (APL).
* AML with normal karyotype and bZIP intramolecular mutations in CEBPA.
* ≥ CR2 status.
* Patients strongly demanding transplantation, and with indications for transplantation but not eligible for transplantation.
* Uncontrolled active infection.
* Severe organ dysfunction.
* Pregnancy.
* Unwillingness to undergo interferon treatment.
* Previous hyperthyroidism or hypothyroidism.
* Participation in other clinical trials within one month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-month negative conversion of MRD | Participants will be followed for a minimum of 2 years until the last enrolled participants was followed up for at least 2 years.
  MFC-MRD or RT-PCR genes (AML1-ETO, NPM1, and CBFb-MYH11) transition from positive to negative.

SECONDARY OUTCOMES:
CIR | Participants will be followed for a minimum of 2 years until the last enrolled participants was followed up for at least 2 years.
  The number of patients with relapse calculated from the randomization time to the last follow-up time.
EFS | Participants will be followed for a minimum of 2 years until the last enrolled participants was followed up for at least 2 years.
  Events include treatment failure (MRD positivity or molecular progression), relapse, or death from any cause.
OS | Participants will be followed for a minimum of 2 years until the last enrolled participants was followed up for at least 2 years.
  calculated from randomization time to the time of death or the last follow-up time.
Treatment-related Safety Indicators | Participants will be followed for a minimum of 2 years until the last enrolled participants was followed up for at least 2 years.
  Mainly include hematologic toxicity and liver toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China